CLINICAL TRIAL: NCT06933043
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous NAV-240 in Healthy Participants
Brief Title: A Study on the Safety, Tolerability, Bioavailability and Mechanism of Action of Intravenous NAV-240 in Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Southern Star Research (Industry)
Collaborators: Navigator Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAV-240-02
Record Dates: First submitted 2025-03-31; First posted 2025-04-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: health volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NAV-240 (Experimental): Participants will be enrolled in 1 of 3 multiple ascending dose cohorts. Six participants in each cohort will receive NAV-240.
  Interventions: Drug: NAV-240
- Placebo to match NAV-240 (Placebo Comparator): In each multiple ascending dose cohort, 2 participants will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NAV-240 — Three doses of intravenous (IV) low dose, medium dose or high dose NAV-240 will be administered to participants.
  Arms: NAV-240
Drug: Placebo — Three doses of matching placebo will be administered to participants.
  Arms: Placebo to match NAV-240

SUMMARY:
The goal of this clinical trial is to assess initial safety/tolerability of multiple doses of drug NAV-240. It will also learn about the profile and immunogenicity of drug NAV-240. The main question it aims to answer is:

• What medical problems do participants have when taking multiple doses of drug NAV-240? Researchers will compare drug NAV-240 to a placebo (a look-alike substance that contains no drug) to see if any medical problems participants have differ between those taking drug NAV-240 and those taking placebo.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, multiple ascending dose (MAD) study will evaluate the safety, tolerability, pharmacokinetics (PK)/pharmacodynamics (PD), and immunogenicity of NAV-240.

ELIGIBILITY:
Selected Inclusion Criteria:

* Male and female participants 18 - 65 years of age
* Medically healthy, in the opinion of the Investigator, with no clinically significant findings on medical history, physical examination, vital signs, or electrocardiograms (ECGs) at Screening, and/or before administration of the initial dose of study drug.
* Participants must have clinical laboratory values within normal ranges of upper limit of normal (ULN) as specified by the testing laboratory, unless deemed not clinically significant (NCS) by the Investigator.
* Body mass index (BMI) 18 to ≤35 kg/m2 at Screening.
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1.
* Female participants of childbearing potential who are sexually active with a male partner of reproductive potential must agree to the use highly effective method of contraception established from at least 28 days prior to screening until at least 90 days after study drug dosing.
* Male participants with female partners who are of reproductive potential must agree to the use of a male condom PLUS a highly effective, method of contraception for the duration of the study, and for at least 90 days after study drug dosing. Male healthy participants also must agree to refrain from sperm donation during the study and for at least 90 days after study drug dosing. Note: Males who are surgically sterile (i.e., documented successful vasectomy) will also be required to use a male condom. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.
* Participants must provide signed informed consent prior to study entry and have the ability and willingness to attend and comply with the necessary visits at the study site. They must also receive a copy of the fully executed informed consent document.

Selected Exclusion Criteria:

* A relevant history of severe respiratory disease that required treatment and/or follow up under the direction of a physician.
* Any neurological, psychiatric, vascular, or system disorder that could also affect the evaluation of disease activity assessments.
* Any other significant acute or chronic medical illness that, in the opinion of the Investigator, would impact the participant's ability to complete all study requirements or that might impact the assessment of study data, or the participant has had a clinically significant illness within 30 days prior to study drug dosing per the Investigator's discretion.
* History of alcoholism or drug abuse within the prior 2 years.
* Acute COVID infection (within three months of Screening) or long COVID.
* A history and/or current presence of a clinically significant atopic allergy, hypersensitivity, or allergic reactions.
* Known or suspected clinically relevant drug hypersensitivity to any components of the test and reference investigational product formulation or comparable drugs.
* A history of any infection requiring hospitalization, IV or oral antibiotics, or as otherwise judged clinically significant, within the 3 months prior to Screening, or an opportunistic infection within the past 12 months, or ongoing infection including chronic viral disease.
* A positive test result for drugs of abuse, cotinine, or alcohol at Screening and on Day -1.
* Active tuberculosis (TB) or a history of TB, or a positive TB blood test at Screening.
* Systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg confirmed by repeat.
* Abnormalities on 12-lead echocardiogram (ECG) prior to study drug dosing, confirmed by repeat.
* All prescription and over-the-counter medications (including vitamins and dietary or herbal supplements), except for contraceptives and acetaminophen, as needed, are prohibited within 7 days prior to the first study drug administration and throughout the treatment period of the study.
* Received vaccines (whether live, attenuated, or killed/inactivated) within 4 weeks prior to Day 1 or is planning to receive any vaccine over the course of the study. Note, influenza vaccines (inactivated) will be allowed during the study.
* Received anti-TNF therapy in the past, confirmed by participant and Investigator.
* Receipt of any investigational drug within 30 days prior to Screening or 5 half-lives, whichever is longer.
* Females who are pregnant or breastfeeding.
* Active cigarette smoker or has regularly used nicotine or nicotine-containing products
* Any reason which, in the opinion of the Investigator, would prevent the healthy participant from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Presence and severity of any treatment-emergent adverse events (TEAEs) and Serious Adverse Events (SAEs) | Through 6 weeks after last dose of study drug.
  Incidence, nature, and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetics parameter - maximum observed concentration (Cmax) | Through to Day 99.
  Maximum observed concentration of the study drug in serum will be analyzed for all participants
Pharmacokinetics parameter - Time for maximum observed Concentration (Tmax) | Through to Day 99.
  Serum PK Tmax will be analyzed for all participants
Pharmacokinetics parameter - Area under the curve (AUC) | Through to Day 99.
  Area under the curve of the study drug in serum will be analyzed for all participants.
Pharmacokinetics parameter - Volume of distribution (Vz) | Through to Day 99.
  Volume of distribution of the study drug in serum will be analyzed for all participants.
Immunogenicity of study drug - Anti-Drug Antibodies (ADAs) | Through to Day 99.
  Serum Anti-Drug Antibodies will be analyzed for all participants

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Brisbane, Queensland, Australia